CLINICAL TRIAL: NCT01827982
Title: A Double-Blind, Placebo-Controlled, Randomized, Single-Ascending Dose Study To Investigate the Safety, Tolerability and Pharmacokinetics of JNJ-54861911 in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of JNJ-54861911 in Healthy Volunteers Compared With Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR101083; 2013-000215-24 (EudraCT Number)
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Healthy; Safety; Tolerability; Pharmacokinetic; Alzheimer's Disease; JNJ-54861911
MeSH Terms: conditions — Alzheimer Disease | interventions — atabecestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Part 1 - Cohort 1: JNJ-54861911 1 mg (Experimental): Following each dose level the observed safety and tolerability profile will be evaluated. The dose will be escalated only if the observed safety and tolerability profile is acceptable.
  Interventions: Drug: JNJ-54861911 1mg
- Part 1 - Cohort 2: JNJ-54861911 3 mg (Experimental)
  Interventions: Drug: JNJ-54861911 3 mg
- Part 1 - Cohort 3: JNJ-54861911 9 mg (Experimental)
  Interventions: Drug: JNJ-54861911 9 mg
- Part 2 - Cohort 4: JNJ-54861911 9 mg (Experimental)
  Interventions: Drug: JNJ-54861911 9 mg
- Part 2 - Cohort 5: JNJ-54861911 27 mg (Experimental)
  Interventions: Drug: JNJ-54861911 27 mg
- Part 2 - Cohort 6: JNJ-54861911 81 mg (Experimental)
  Interventions: Drug: JNJ-54861911 81 mg
- Part 2 - Cohort 7: JNJ-54861911 160 mg (Experimental)
  Interventions: Drug: JNJ-54861911 160 mg
- Part 3 - Cohort 8: JNJ-54861911 (dose to be determined [tbd]) (Experimental)
  Interventions: Drug: JNJ-54861911 tbd
- Parts 1 through 3 - Placebo (Placebo Comparator): Participants in each cohort will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-54861911 1mg — JNJ-54861911 1 mg will be administered as a single oral dose after an overnight fast of at least 10 hours.
  Arms: Part 1 - Cohort 1: JNJ-54861911 1 mg
Drug: JNJ-54861911 3 mg — JNJ-54861911 3 mg will be administered as a single oral dose.
  Arms: Part 1 - Cohort 2: JNJ-54861911 3 mg
Drug: JNJ-54861911 9 mg — JNJ-54861911 9 mg will be administered as a single oral dose.
  Arms: Part 1 - Cohort 3: JNJ-54861911 9 mg
Drug: JNJ-54861911 27 mg — JNJ-54861911 27 mg will be administered as a single oral dose.
  Arms: Part 2 - Cohort 5: JNJ-54861911 27 mg
Drug: JNJ-54861911 81 mg — JNJ-54861911 81 mg will be administered as a single oral dose.
  Arms: Part 2 - Cohort 6: JNJ-54861911 81 mg
Drug: JNJ-54861911 160 mg — JNJ-54861911 160 mg will be administered as a single oral dose.
  Arms: Part 2 - Cohort 7: JNJ-54861911 160 mg
Drug: JNJ-54861911 tbd — The dose of JNJ-54861911 will be derived from the results obtained in Parts 1 and 2.
  Arms: Part 3 - Cohort 8: JNJ-54861911 (dose to be determined [tbd])
Drug: JNJ-54861911 9 mg — Study drug will be administered after an overnight fast of at least 10 hours and within 120 minutes after placement of the spinal catheter.
  Arms: Part 2 - Cohort 4: JNJ-54861911 9 mg
Drug: Placebo — Matching placebo will be given as a single oral dose.
  Arms: Parts 1 through 3 - Placebo

SUMMARY:
The purpose of this study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of JNJ-54861911 which is currently being developed for the treatment of Alzheimer's Disease.

DETAILED DESCRIPTION:
This study is a first-in-human, double-blind (neither investigator nor participant knows which treatment the participant receives), randomized (participants are assigned different treatments based on chance), placebo-controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), single-ascending dose study. The study is designed to evaluate the safety (side effects), tolerability and pharmacokinetics (how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time, ie, what the body does to the drug), and pharmacodynamics (what the drug does to the body) of JNJ-54861911 which is currently being developed for the treatment of Alzheimer's Disease.

The study population will consist of approximately 64 healthy participants divided among approximately 8 cohorts (small groups). Each cohort will have 8 participants.

For all participants the study will consist of 3 phases: a screening phase (between 28 and 2 days prior to the first dose administration), a double-blind treatment phase, and a follow-up examination (within 7 to 14 days after last dose administration). Participants who successfully complete the screening examination and are considered eligible to participate will be admitted to the clinical unit on Day -1 before administration of the study drug and will remain in the unit until the evening of Day 3.

The double-blind treatment phase will consist of three parts: Part 1 (Cohorts 1 to 3) is a single ascending dose part in young healthy male participants, between 18 and 54 years of age. Part 2 (Cohorts 4 to 7) is a single-ascending dose part in elderly male and female participants between 55 and 75 years of age including continuous cerebrospinal fluid (CSF) sampling. Within Parts 1 and 2 of the study, participants will be randomized (assigned by chance) to treatment with JNJ-54861911 (n=6/cohort) or matching placebo (n=2/cohort). Following each dose level, the observed safety and tolerability profile will be evaluated. If no side effects are observed and the pharmacokinetic data are roughly in line with predicted safe values, the dose will be escalated. Each participant of the next cohort will be given a higher dose of JNJ-54861911. As a general safety precaution for a first-in-human study, all dose administrations in Part 1, Cohort 1 and all further cohorts will be staggered.

Part 1 of the study will primarily focus on determining safety and tolerability of JNJ-54861911 after single ascending dose administrations and understanding the primary pharmacokinetic characteristics of JNJ-54861911. In addition possible pharmacodynamic effects of JNJ-54861911 on plasma amyloid beta (Aβ) levels will be explored. The primary focus of Part 2 will be determining the maximal tolerated dose level of JNJ-54861911 or determine the safety and tolerability at the maximum feasible exposure level, whichever is reached first in healthy elderly participants. In addition the reduction in CSF Aβ over 36 hours post single dose administration of JNJ-54861911 will be explored. Planned doses will be 1 mg, 3 mg, 9 mg, 27 mg, 81 mg, and 160 mg of JNJ- 54861911 or matching placebo, administered as a single oral dose. The starting dose of JNJ-54861911 in Part 2 will be the dose level tested in Part 1 found to be safe and well tolerated, and that is expected to reduce CSF Aβ by 20 percent or more. The initial dose tested in Part 2 will not be higher than the doses tested in Part 1.

Part 3 (Cohort 8) of the study will evaluate the effect of food on how JNJ-54861911 is absorbed, distributed within the body, and removed from the body. One single dose of JNJ-54861911 or matching placebo will be tested after consumption of a high fat breakfast. The dose of JNJ-54861911 tested in this part will be derived from the results obtained in Parts 1 and 2. Part 3 may be performed in parallel with Part 1 or 2 of the study. Depending on the pharmacokinetic properties and safety and tolerability profile of JNJ-54861911, young or elderly healthy participants may be recruited for this part. In addition male participants enrolled in Part 1 or Part 2 may also be enrolled for Part 3.

Participants will be discharged from the clinical unit after the last study assessment on Day 3 has been obtained. Participants will only be discharged if in the opinion of the investigator it is safe for the participants to be discharged. The participant will return to the clinical unit on Day 4 (72 h post dose) and Day 5 (96 h post dose) for plasma PK sampling. Safety assessments will be performed throughout the study. The maximal study duration for a participant will not exceed 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Must adhere to required contraception during and for 3 months after study

Specific Inclusion Criteria for Part 1:

* Body mass index between 18 and 30 kg/m2
* Male volunteers, between 18 and 54 years of age, inclusive

Specific Inclusion Criteria for Part 2:

* Body mass index between 18 and 32 kg/m2
* Women must be postmenopausal, permanently sterilized or otherwise be incapable of pregnancy
* Healthy male or female volunteers, between 55 and 75 years of age, inclusive

Specific Inclusion Criteria for Part 3:

* Male volunteers
* If participated in Parts 1 or 2, specific inclusion criteria for Part 1 (young) or Part 2 (elderly) may apply

Exclusion Criteria:

* Clinically significant medical or psychiatric illness
* Alcohol or substance abuse; excessive nicotine or caffeine use
* Recently received an investigational drug, vaccine, or invasive medical device
* Unable to abide by protocol restrictions on use of other medications
* History or family history of spontaneous, prolonged or severe bleeding of unclear origin or of blood clotting
* Current anemia

Specific Exclusion Criteria for Part 2:

* History of lower back pain or scoliosis and/or major (lumbar) back surgery
* Allergic to local anesthetics and/or iodine
* Increased intracranial pressure based on fundoscopy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of JNJ-54861911 | Up to 96 hours
  The maximal tolerated dose (MTD) after single dose administration of JNJ-54861911 or the safety and tolerability at the maximum feasible dose level, whichever is reached first

SECONDARY OUTCOMES:
Maximum observed plasma/cerebrospinal fluid (CSF) concentration (Cmax) of JNJ-54861911 | Up to 96 hours post-dose
  Cmax is observed maximum plasma concentration of study drug, taken directly from the plasma concentration-time profile
Time to reach maximum observed plasma/CSF concentration of JNJ-54861911 | Up to 96 hours post-dose
  Time when Cmax is observed, taken directly from the plasma concentration-time profile
Area under the plasma/CSF concentration-time curve (AUC) from time 0 to t hours of JNJ-54861911 | Up to 96 hours post-dose
  The AUC (0 to t hours) is area under the plasma concentration-time curve from time 0 to t hours after dosing; t is time of the quantifiable concentration Clast
Half-life of JNJ-54861911 | Up to 96 hours post-dose
  Defined as 0.693/elimination rate constant
Amyloid Beta profile in cerebrospinal fluid (CSF) | Up to 36 hours post-dose
Elimination rate constant | Up to 96 hours post-dose
  Elimination rate constant is determined by linear regression of the terminal points of the ln-linear plasma/CSF concentration-time curve
Area under the plasma/CSF concentration-time curve from time 0 to infinity of JNJ-54861911 | Up to 96 hours post-dose
  The AUC (0 to infinity) is area under the plasma concentration-time curve from time 0 to t hours extrapolated to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Antwerp, Belgium